CLINICAL TRIAL: NCT01017926
Title: An Open, Two Period, Two Treatment, Two Sequence, Crossed, Randomized, Single-Dose Study Of Two Oral Preparations Containing 0.25 Mg Of Triazolam (Halcion, Pharmacia & Upjohn S.A. De C.V. Vs. Product Made By Pfizer Pharmaceuticals LLC) In Healthy Volunteers Under Fasting Conditions
Brief Title: Triazolam Trial In Healthy Subjects To Compare Bioavailability Between Formulations Of Triazolam To Determine Their Bioequivalence In Terms Of Rate And Magnitude Of Absorption
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Collaborators: Investigación Farmacológica y Biofarmacéutica (Unknown)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer, Inc.
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: A6781002
Record Dates: First submitted 2009-11-20; First posted 2009-11-23 (Estimated); Last update posted 2016-04-06 (Estimated); Status verified 2016-04

CONDITIONS: Healthy Volunteers
Keywords: Triazolam bioequivalence
MeSH Terms: interventions — Triazolam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Triazolam Reference Arm (Active Comparator): There will be a clearance period of at least 3 days between the two phases of the study.
  Interventions: Drug: Triazolam
- Triazolam Trial Arm (Experimental)
  Interventions: Drug: Triazolam

INTERVENTIONS:
Drug: Triazolam — Tablets, 0.25 mg, single-dose, 1 period of 3 three days.
  Arms: Triazolam Reference Arm
Drug: Triazolam — Tablets, 0.25 mg, single-dose, 1 period of 3 three days.
  Arms: Triazolam Trial Arm

SUMMARY:
The purpose of this study is to compare the bioavailability of two oral formulations of Triazolam in healthy volunteers, in order to determine that they are bioequivalent.

DETAILED DESCRIPTION:
The bioequivalence trial of triazolam is due to change in manufacture site.

ELIGIBILITY:
Inclusion Criteria:

* Only healthy volunteers, between the ages of 18 and 40 years, will be included.
* Subjects' body mass index must be between 19-27.
* Volunteers must be in good health, as determined by the results of a complete clinical history prepared by doctors at the clinical research site and laboratory tests performed at certified clinical laboratories.
* Volunteers must agree to use at least two birth control methods (except hormonal contraceptives) from the first dose of the study drug and for up to 28 days after the last dose. (acceptable methods are surgically definitive sterilization, menopause, barrier methods such as condoms and diaphragm, and spermicidal gels/foams)
* The limits of variation permitted within normality at the screening visit will be: blood pressure (seated) 90 to 130 mm Hg systolic and 60 to 90 mm Hg diastolic, heart rate between 55 and 100 beats per minute and respiratory rate between 14 and 20 respirations per minute.
* The laboratory and cabinet tests required to include subjects in the studio will be: 1) Hematology: hemoglobin, hematocrit, total white blood cell count with differential, and platelet count, 2) 27-element blood chemistry, 3) Markers for hepatitis B and C. 4) Detection of HIV, 5) General urinalysis, 6) Drug abuse test in both study periods, 7) Qualitative pregnancy test in both study periods (if applicable) , 8) Electrocardiogram. (pre-screening/recruitment)

Exclusion Criteria:

* Subjects in whom any alteration is detected in their vital signs recorded at the screening of volunteers.
* Volunteers who fail to comply with the established criteria for inclusion.
* Volunteers with antecedents of cardiovascular, renal, hepatic, muscular, metabolic, and gastrointestinal disorders, including constipation; neurological, endocrine, and hematopoietic disorders; or any kind of anemia, asthma, mental illness, or other organic abnormalities, as well as those who have suffered a muscular traumatism within 21 days before the study.
* Volunteers who require any medication over the course of the study, aside from the drug being studied.
* Volunteers with antecedents of dyspepsia, gastritis, esophagitis, and duodenal or gastric ulcers.
* Volunteers who have been exposed to known hepatic enzyme inductors or inhibitors or have taken potentially toxic drugs within 30 days before the start of the study.
* Volunteers who have received any medication within 14 days or 5 half lives (whichever is longer) before the start of the study.
* Volunteers who have been hospitalized for any problem within seven months before the start of the study.
* Subjects who have received investigational drugs within 60 days prior to the study.
* Subjects allergic to any antibiotic and/or non-steroidal antiinflammatory analgesics.
* Subjects who have consumed alcohol or xanthine containing beverages (coffee, tea, cocoa, chocolate, mate, colas) or have consumed charcoal broiled foods or grapefruit juice within one week before the start of the study and until the last sample is taken.
* Subjects who have donated or lost 450 mL or more of blood within 60 days before the start of the study.
* History of regular consumption of alcohol exceeding 14 drinks/week (1 drink = 5 ounces (150 mL) of wine or 12 ounces (360 mL) of beer or 1.5 ounces (45 mL) of liquor within 6 months before the screening visit.
* Excessive use of products containing tobacco or nicotine, equivalent to 5 cigarettes per day.
* Female volunteers with positive results on the pregnancy test or in lactation.
* Volunteers who require a special diet for any reason, for example vegetarians.
* Disability of any kind that prevents the volunteer from understanding the nature, purpose, and potential consequences of the study.
* Evidence of an uncooperative attitude during the study.
* Female volunteers in lactation.
* Female volunteers who receive oral contraceptives

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2010-08; Primary Completion 2010-09 (Estimated); Study Completion 2010-09 (Estimated)

PRIMARY OUTCOMES:
Establish Cmax, Tmax, elimination half life, area below the curve from zero to t, and area below the curve from zero to infinity (ABC 0-∞) of the two formulations of Triazolam in tablets | Day 1 and two after dosage is taken
Statistically compare the bioavailability of the pharmaceutical formulations of Triazolam studied, to establish or rule out the existence of bioequivalence | Six to eight weeks after completing the study, a final report will be prepared.

SECONDARY OUTCOMES:
Investigate the safety of both preparations based on the record of adverse events on completing both study periods | Up to 3 days after the 2nd period

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6781002